CLINICAL TRIAL: NCT05235672
Title: Detection of Latent Autoimmune Diabetes in Adults, Clinical and Metabolic Profile in Patients Treated at the Diabetes Clinic in a Hospital in the Mexican Southeast.
Brief Title: Detection of LADA in a Hospital in the Mexican Southeast
Acronym: LADA patients
Status: Completed | Type: Observational
Sponsor: Universidad Juárez Autónoma de Tabasco (Other)
Responsible Party: Principal Investigator, ISELA ESTHER JUAREZ-ROJOP Ph.D., Professor, Universidad Juárez Autónoma de Tabasco
Other Study IDs: LADA-DACS
Record Dates: First submitted 2022-01-25; First posted 2022-02-11 (Actual); Last update posted 2022-02-11 (Actual); Status verified 2022-02

CONDITIONS: Latent Autoimmune Diabetes
Keywords: LADA; GADA; Mexican population

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patients with Latent Autoimmune Diabetes in Adults (LADA) show autoantibodies that indicate an autoimmune pathogenesis. Glutamic acid decarboxylase autoantibodies (GADA) are most prevalent islet autoantibodies in European patients with LADA. In this sense, it is considered that it is sufficient to determine GADA to identify subjects with LADA from patients with T2D for research purposes. Therefore, the aim was to investigated the presence of GADA in serum of subjects with T2D and its relationship with clinical criteria, metabolic control, drug treatment, and diabetes complications to identify possible patients with LADA in a hospital in southeastern Mexico is worthwhile.

The sample was recruited at the Diabetes Clinic of the Regional Hospital of High Specialty "Dr. Gustavo A. Rovirosa Pérez", in the period from January 2020 to May 2021. The diagnosis was based in accordance with World Health Organization (WHO, 1999) criteria. Inclusion criteria: 1) patients previously diagnosed with T2D, 2) absence of insulin requirement for at least 6 months after diagnosis, 3) > 30 and < 50 years old at diabetes diagnosis, 4) BMI < 40 kg/m2, 5) subjects who agreed to participate in the study and signed the informed consent before the interview.

Serum GADA and other biochemical concentrations were determined by an enzymatic immunoassay method (Human Anti-Glutamic Acid Decarboxylase ELISA Kit; MyBioSource).

ELIGIBILITY:
Inclusion Criteria:

* patients previously diagnosed with T2D,
* absence of insulin requirement for at least 6 months after diagnosis,
* > 30 and < 50 years old at diabetes diagnosis,
* BMI < 40 kg/m2,
* subjects who agreed to participate in the study and signed the informed consent before the interview.

Exclusion Criteria:

• patients with other types of diabetes, and subjects who did not agree to participate.

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Subjects were initially diagnosed and received pharmacological treatment for T2D. In addition, these patients presented clinical and biochemical characteristics both of T1D and T2D, progressing to insulin dependency. Such individuals were invited to participate in the study. An endocrinologist diagnosed and evaluated all these patients.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2021-01-30 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
GADA in serum of subjects with T2D | May 2021
  Serum GADA concentrations were determined by an enzymatic immunoassay method in subjects with T2D

CONTACTS AND LOCATIONS:
Locations (1):
- Isela Esther Juarez Rojop, Villahermosa, Tabasco, Mexico